CLINICAL TRIAL: NCT00933894
Title: A Phase I, Open-label, Randomized, Crossover Trial in 16 Healthy Subjects to Investigate the Potential Pharmacokinetic Interaction Between Telaprevir and Escitalopram at Steady-state
Brief Title: VX-950-TiDP24-C133 - A Phase I Study Investigating the Interaction Between Telaprevir and Escitalopram
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec BVBA (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016303
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Hepatitis C
Keywords: VX-950-TiDP24-C133; VX-950-C133; VX950; HCV; telaprevir; escitalopram
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Escitalopram

INTERVENTIONS:
Drug: Telaprevir; Escitalopram

SUMMARY:
The purpose of this study is to investigate the effect of steady-state telaprevir (TVR) 750 mg q8h (3 times a day, every 8 hours) on the steady-state pharmacokinetics of escitalopram 10 mg q.d. (once a day), and vice versa. Steady state is a term which means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. TVR is being investigated for the treatment of chronic hepatitis C virus (HCV) infection. Pharmacokinetics (pk) means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body.

DETAILED DESCRIPTION:
Telaprevir is being investigated for treatment of chronic HCV infection, in combination with Peg-IFN (pegylated interferon) and RBV (ribavirin). Peg-IFN plus RBV are currently an accepted methode for treating HCV. Treatment with Peg-IFN plus RBV for HCV infection is associated with a high rate of depression. The results of this study will provide dosing recommendations for coadministration of Telaprevir (TVR) and escitalopram in HCV-infected patients. This is a Phase I, open-label (both participant and investigator know the name of the medication), randomized (study medication assigned by chance), crossover trial in 16 healthy participants to investigate the pharmacokinetic interaction between escitalopram and TVR, both at steady state. Steady state is a term which means that the drug has been given long enough so that the plasma concentrations will remain the same with each subsequent dose. The participants will receive two treatments (treatment A-B or treatment B-A) in a randomized order. In Treatment A, participants will receive escitalopram 10 mg once daily (q.d.) for 7 days. In Treatment B, participants will receive TVR 750 mg every 8 hours (q8h) for 14 days, with coadministration of escitalopram 10 mg q.d. from Day 8 to Day 14. There will be a washout period (a period where no treatment will be taken in view of having all the medication eliminated from the body before starting a new treatment) of at least 14 days between last intake of study medication in one session and first intake of study medication in the subsequent session. All study medication will be taken with food. Escitalopram will be taken once daily in the morning. During coadministration of TVR and escitalopram, the first dose of TVR should be taken together with escitalopram in the morning. Pharmacokinetic profiles of the two compounds will be measured through blood samples taken at regular intervals during the study and safety and tolerability will be assessed during the study period and in follow-up. Safety and tolerability evaluations will be recorded at regular intervals throughout the trial period. Blood and urine samples, electrocardiogram (ECG) and vital signs (blood pressure and hart rate) will be taken at screening, before medication intake on days 1 and 7 in each session and on day 14 in treatment B and at the 2 follow up visits at 5-7 and 30-32 days after last dose of drug in the last session. A physical examination will be performed at screening, on day before first medication intake in each session and during the 2 follow up visits. Participants in Treatment A will receive oral escitalopram 10 mg once daily for 7 days and in Treatment B participants will receive TVR 750 mg q8h from Day 1 to Day 14, with coadministration of escitalopram 10 mg q.d. from Day 8 to Day 14.

ELIGIBILITY:
Inclusion Criteria:

* Females should be post-menopausal for at least 2 years (amenorrheal for at least 3 years), or have undergone tubal ligation (or other permanent birth control methods), or hysterectomy (total), or oophorectomy (bilateral), and should not be breastfeeding
* Nonsmoking or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months before study screening
* Body mass index (BMI, weight in kg divided by the square of height in meters) of 18 to 30 kg/m2, extremes included, at study screening
* normal 12-lead ECG at screening
* Healthy on the basis of a physical examination, medical history, vital signs, and the results of blood chemistry, hematological and coagulation tests and urinalysis carried out at screening

Exclusion Criteria:

* Participants should stop any short-duration courses of prescription medication at least 14 days before first intake of study medication, potential participants should not stop any chronic, prescribed medication being taken at the direction of a physician, without obtaining agreement from that physician
* Participants should stop over-the-counter medications on the date of the screening visit but no less than 7 days prior to the first administration of study medication, potential participants should not stop any chronic, over-the-counter medication being taken at the direction of a physician, without obtaining agreement from that physician
* Consumption of more than 2 units of alcoholic beverages per day or more than 14 units per week (1 unit of alcohol equals 1 glass [285 mL] of beer, 1 glass [125 mL] of wine, 25 mL shot of 40% spirit) from 14 days before the first intake of study medication until completion of the pharmacokinetic sampling in the last treatment session
* Participants may not consume any alcohol 72 hours before or after study drug administration
* Positive test for any of the following infectious disease tests: hepatitis A infection (confirmed by hepatitis A antibody IgM), hepatitis B antigen (HBsAg), hepatitis C virus antibody (HCVAb), human immunodeficiency virus 1 antibody (HIV1Ab), or human immunodeficiency virus 2 antibody (HIV2Ab)
* Male participants with female partners that are planning to become pregnant during the study or within 90 days of the last dose of study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To investigate the effect at steady-state of TVR 750 mg q8h on the steady-state pharmacokinetics of escitalopram 10 mg q.d. in healthy participants and vica versa. | pk profiles of TVR will be measured up to 8 hours after intake of the morning dose on Day 7 and 14 of Treatment B. Pharmacokinetic profiles of escitalopram will be measured up to 24 hours postdose on Day 7of Treatment A and Day 14 of Treatment B.

SECONDARY OUTCOMES:
The short-term safety and tolerability of coadministration of TVR and escitalopram in healthy participants | This will be determined throughout the study; at all study visits

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec-Virco Virology BVBA Clinical Trial, Study Director — Tibotec BVBA